CLINICAL TRIAL: NCT04781673
Title: A Prospective, Randomized, Single-Blinded Trial of Ketamine Versus Lidocaine Infusions for Multimodal Pain Management in Traumatic Rib Fracture Patients
Brief Title: Ketamine vs Lidocaine in Traumatic Rib Fractures
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brittany Hoyte (Other)
Responsible Party: Sponsor-Investigator, Brittany Hoyte, Principal Investigator, Corewell Health West
Organization: Corewell Health West (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-508
Record Dates: First submitted 2021-02-22; First posted 2021-03-04 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Rib Fractures; Rib Fracture Multiple; Rib Trauma
Keywords: Lidocaine; Ketamine; Rib Fracture; Traumatic Rib Fracture
MeSH Terms: conditions — Rib Fractures | interventions — Ketamine; Lidocaine

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Trial, Single-blinded
Who Masked: Participant
Masking Description: Medication infusion and medication IV bag will be covered with brown protect from light bag
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketamine (Active Comparator): Infusion initiation: 0.1 mg/kg/hr Max: 0.3 mg/kg/hr Recommended titration: 0.1 mg/kg/hr* as needed every 4 hours based on pain scores ≥5 and physician order
  Dosing will be based on patient actual body weight (ABW) recorded as dosing weight on time of hospital admission.
  Interventions: Drug: Ketamine
- Lidocaine (Active Comparator): Infusion initiation: 1 mg/kg/hr Max: 2 mg/kg/hr Recommended titration:0.25 mg/kg/hr* as needed every 4 hours based on pain scores ≥5 and physician order
  Dosing will be based on patient actual body weight (ABW) recorded as dosing weight on time of hospital admission.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Ketamine — Will receive titratable infusion.
  Other Names: Ketalar
  Arms: Ketamine
Drug: Lidocaine — Will receive titratable infusion, will have daily lidocaine level labs drawn daily.
  Other Names: Xylocaine
  Arms: Lidocaine

SUMMARY:
Rib fractures continue to be a common occurrence in trauma patients of all ages. Traumatic rib fractures can cause severe pain in patients and lead to shallow breathing and further complications such as the need for mechanical ventilation, hospital or ventilator associated pneumonia, atelectasis, and acute respiratory distress syndrome. Effective multimodal pain management is needed to optimize a patient's respiratory status and can also play a role in early mobility, less pulmonary complications, shorter ICU and hospital length of stay, and decreased mortality. Current multimodal pain management options include opioids, muscle relaxants, gabapentin, acetaminophen, nonsteroidal anti-inflammatory drugs, and various regional/neuraxial anesthesia techniques. Both ketamine and lidocaine infusions for pain control have also been shown in studies to be safe and effective, with the benefit of minimizing the use of opioids. However, there have been very few studies that have used ketamine or lidocaine infusions for pain control specifically in patients with traumatic rib fractures. Therefore, the purpose of this study is to evaluate ketamine versus lidocaine infusions as an adjunctive therapy to reduce opioid consumption in the first 72 hours in patients with multiple traumatic rib fractures.

DETAILED DESCRIPTION:
Effective pain control plays a key role is optimizing a patient's respiratory status after suffering multiple rib fractures. Using multimodal pain management techniques and optimizing a patient's pain control regimen helps to minimize the complications associated with rib fractures, such as pneumonia and the need for mechanical ventilation. The benefit of using opioid-sparing options such as ketamine or lidocaine infusions would be to avoid the side effects associated with opioids, which include delirium, constipation, and depressed respiratory drive.

Ketamine and lidocaine infusions are both medications that have been used in numerous studies to effectively treat post-operative pain. Low dose ketamine infusions have also recently been shown to be a safe and effective adjunct option to help reduce pain scores and decrease opioid use in patients with traumatic rib fractures. Currently there is no published studies to assess lidocaine's effectiveness to reduce pain scores and opioid use in traumatic rib fracture patients. There is also only one study to date that has directly compared ketamine to lidocaine infusions for pain control. This study occurred in 60 patients undergoing elective nephrectomy and evaluated three 24-hour infusion groups: ketamine, lidocaine, or placebo. The primary outcome showed that both ketamine and lidocaine infusions significantly reduced 24-hour OME compared to placebo (33% ketamine, 42% lidocaine) and decreased overall pain scores.

This trial is a single center, prospective, randomized trial of adult patients with ≥ 3 traumatic rib fractures admitted to a Level 1 trauma center at Spectrum Health Butterworth Hospital. As part of the current rib fracture protocol all patients will receive the standard multimodal pain regimen at the investigator's institution, including acetaminophen, NSAIDS, muscle relaxants and gabapentin. Currently ketamine infusions and regional/neuraxial anesthesia techniques are added if the standard multimodal pain regimen is insufficient. Lidocaine infusions have also been used at the institution for post-surgical pain control to minimize opioid use. The objective of the study will be to compare ketamine versus lidocaine infusions on the effectiveness to optimize pain control as well as minimize the use of opioids in patients with traumatic rib fractures.

If consent is obtained the patient will be randomized 1:1 to receive either a ketamine or lidocaine infusion for pain control, along with standard of care, using a pre-designed randomization schedule. Patients must be enrolled within 16 hours of hospital admission and are expected to remain on the infusion for a minimum of 24 hours. The duration, titration, and stopping of study drug will be dependent on the progress of the patient's overall pain status and provider decision, with data being included for the study medication for up to 72 hours. If patients require surgery at any time the study medication will not be held unless signs of adverse events occur. Patients who are unable to remain on the study infusion or have a regional/neuraxial anesthetic placed before the 24-hour mark (decided based on the Trauma and Surgical Intensive Care Unit services) will be considered a screen fail and no data will be contributed to the study, however, the screen fail will be documented. If a patient is unable to remain on infusion or has a regional/neuraxial anesthetic placed ≥ 24 hours, their data will be included up until that point and analyzed. Adverse event and serious adverse events will be monitored throughout the entire study period, with continuous cardiac telemetry being required in both study groups and daily lidocaine levels drawn in the lidocaine group.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years old
2. ≥ 3 traumatic blunt rib fractures
3. Enrollment within 16 hours of being admitted to the hospital
4. Patients whom in the investigator's clinical judgement, would require escalated pain control regiments in the future and would potentially benefit from participation in this study in terms of pain control.

Exclusion Criteria:

1. Patients receiving any regional/neuraxial anesthetic techniques or ketamine infusion before randomization
2. Adults with diminished decision-making capacity
3. Adults of limited English proficiency/non-English speakers
4. Prisoners
5. Pregnant or breastfeeding women
6. Patient admission weight greater than 120 kg
7. Patients with any of the following medical history:

   1. Active delirium (as defined by Confusion Assessment Method)
   2. Dementia
   3. Psychosis
   4. Glaucoma
   5. Heart block (except with patients with a functioning artificial pacemaker)
   6. Congestive heart failure (ejection fraction <20% recorded in last year)
   7. Adams-Stokes syndrome
   8. Wolff-Parkinson-White Syndrome
8. Patient is unable to communicate with staff for pain assessments at time of enrollment
9. Most recent documented Glasgow Coma Score <15 at the time of study enrollment
10. Severe bradycardia (heart rate <50 bpm based on last vital sign recorded at time of study enrollment)
11. Sustained hypertension (systolic blood pressure >180 mm Hg or diastolic blood pressure >100 mm Hg for at least 3 sets of vital signs in a row prior to study enrollment)
12. Any seizure suspected or identified during hospital admission
13. Patient with active acute coronary syndrome obtained from admission problem list
14. Patients with known hepatic disease or acute liver failure

    a. Acute liver failure on admission defined as either: i. International normalized ratio > 1.5, without being on home anticoagulation ii. Aspartate aminotransferase or Alanine aminotransferase greater than 120 IU/L (3 times upper limit of normal) b. Known hepatic disease defined as past medical history of Child Turcotte Pugh (Child's) score C
15. Patients with a history of end-stage renal disease or admission creatinine clearance (CrCl) ≤30 ml/min

    a. CrCl will be based on Cockcroft-Gault equation from admission labs
16. Use of antiarrhythmic medication therapy prior or during admission

    a. Amiodarone, sotalol, dofetilide, dronedarone, mexilitine
17. Patients with a known allergy/sensitivity to lidocaine or ketamine, amide anesthetics, or components of the solution
18. Patients who, in the investigator's opinion, should not be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Oral Morphine Equivalent - Opioid Usage | 0-24 hours post infusion
  Oral morphine equivalence is a way to track the amount of opioids used by standardizing all opioid utilizations and converting them to daily morphine equivalence in mg.

SECONDARY OUTCOMES:
Visual Analogue Numeric Pain Score | 0-24; 24-48; 48-72 hours post infusion
  Visual Analogue Numeric Pain Score are recorded as a scale of 1-10, with 0 being no pain and 10 as worst imaginable pain. Patient will be asked their pain score every 6 hours.
Oral Morphine Equivalent - Opioid Usage | 24-48; 48-72 hours post infusion
  Oral morphine equivalence is a way to track the amount of opioids used by standardizing all opioid utilizations and converting them to daily morphine equivalence in mg.
Respiratory Failure | 0-30 days post-infusion
  Respiratory failure was defined by need for mechanical intubation
Use of Regional/Neuraxial anesthesia | 0-30 days post infusion
  Measure of regional/neuraxial anesthesia placement rates. Patient would need to be taken off study medication if decision made to place regional/neuraxial anesthetic.
Hospital Length of Stay | Will capture retrospectively after patient's medical discharge
  Total hospital length of stay up to 365 days
Intensive Care Unit Length of stay | Will capture retrospectively after patient's medical discharge
  Total intensive care unit length of stay up to 365 days
Incentive Spirometry | 0-24; 24-48; 48-72 hours post infusion
  Measure of percent improvement in incentive spirometry level from baseline (before infusion). Incentive spirometry levels range from 0-4,000 mL.
Adverse events | 0-72 hours post infusion
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
In-Hospital mortality | Will capture retrospectively after patient's medical discharge
  Patient's death will be recorded if it occurs before discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Corewell Health West, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No